CLINICAL TRIAL: NCT06653504
Title: The CONUS-BRS STUDY: An Observational, Analytical, Cross Sectional Study Investigating the Effects of Conus Branch and Right Ventricular (RV) Branch Occlusion on Surface ECG and Intra-cardiac Electrograms in Patients Undergoing Percutaneous Coronary Intervention (PCI)
Brief Title: The Conus Brugada Syndrome Study
Acronym: Conus-BRS
Status: Completed | Type: Observational
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1 08/12/2016
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Brugada Syndrome
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An observational, analytical, cross sectional study investigating the effects of Conus branch and Right Ventricular (RV) Branch occlusion on surface ECG and intra-cardiac electrograms in patients undergoing percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85
* Patients able and willing to give their written informed consent.
* Planned PCI of a CTO of a right coronary artery
* Planned use of an anchor balloon in the Conus branch or RV branch

Exclusion Criteria:

* Patients considered unsuitable to participate by the research team (e.g., due to medical reasons, laboratory abnormalities, or subject's unwillingness to comply with all study related procedures).
* Patients with a pre-existing, confirmed or possible diagnosis of Brugada Syndrome
* Marked ST elevation or J point elevation on baseline (prior to procedure) ECG in the precordial leads (V1-V3)
* Pregnancy. This will be tested by urine HcG measurement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients aged at least 18 years who have a chronic total occlusion of the RCA with no significant anterior ST elevation prior to an elective CTO procedure.
  2. A Conus branch and or RV branch present to deploy an anchor balloon.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
ECG and/or electrogram changes | During Procedure
  Incidence of ECG changes resembling a Brugada type 1 pattern of coved ST elevation (one of the three Brugada types) specifically significant J point elevation in the precordial leads (V1-V3) and/or electrogram changes on the epicardial and/or endocardial intracardiac traces which will then be compared for differences and evidence of a transmural voltage gradient existing between them.

CONTACTS AND LOCATIONS:
Overall Officials: Pier Lambiase, PhD FRCP FHRS, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom